CLINICAL TRIAL: NCT04435093
Title: Digitalization Playful Module of Motor Function Measure Assessment for Children With Neuromuscular Disorders, MFM-Play Pilot Study.
Acronym: MFM-Play pilot
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0150; 2020-A01752-37 (Other: ID-RCB)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MFM completion
  Interventions: Other: MFM-Play

INTERVENTIONS:
Other: MFM-Play — Neuromuscular patients will complete five items of the MFM (items 18 to 22) either conventionally or using the MFM-Play with 2 different therapists, on the same day. The order of the MFM type completion will be determined by randomization. Both therapists will rate items 18 to 22 blindly.

SUMMARY:
The Motor Function Measure (MFM) is a functional rating scale consisting of 32 items assessing motor functional abilities in a person with neuromuscular disease.

By exploring the potential of digital technologies applied to MFM, for each item completion we want to create digital animations containing different playful and informative scenarios. This digital evolution aims to standardize assessment on the therapist's side, but also to improve acceptance of scale and patient participation.

Despite the modification of the MFM completion by digital animation, the study hypothesis is that the metrological qualities of the scale are retained.

Through the MFM-Play pilot study, the objective is to test 5 items of the MFM-Play scale before carrying out a validation study of the total MFM-Play.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys with a neuromuscular disease
* Aged 6 to 11 years old
* With parental assent

Exclusion Criteria:

* Patients participating to a therapeutic trial
* Patients without compartmental capacities to participate normally to the MFM.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will involve children with a neuromuscular disease, aged 6 to 11 years old
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
MFM scores item 18 to 22 | Day 1
  Level of agreement between the scores obtained during the classic mode and during the MFM-Play mode, completed by two different therapists.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Vincent-Genod, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hospices Civils de Lyon, Bron
  - CHU de Grenoble, La Tronche
  - CHU Saint Etienne, Saint-Etienne